CLINICAL TRIAL: NCT01223547
Title: The Effect of Carbohydrate Counting and Bolus Calculation Using an Electronic Calculator in Carbohydrate Counting-naïve Persons With Non-optimally Treated Type 1 Diabetes
Brief Title: Study of the Effects of Carbohydrate Counting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: The Danish Council for Strategic Research (Other); Medtronic (Industry); Roche Pharma AG (Industry); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Signe Schmidt, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOLUSCAL
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Type 1 Diabetes
Keywords: Carbohydrate counting; Insulin bolus calculation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Participants in this arm continues their usual insulin therapy
- Carb counting (Active Comparator): Participants in this arm are taught carb counting
  Interventions: Other: Education
- Carb counting and bolus calculator (Active Comparator): Participants in this arm are taught carb counting and are provided with an integrated glucose meter and bolus calculator.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Participants are taught the principles of carb counting
  Arms: Carb counting
Other: Education — Participants are taught the principles of carb counting and the use of the integrated glucose meter and bolus calculator.
  Other Names: The integrated glucose meter and bolus calculator: Aviva Expert, Roche
  Arms: Carb counting and bolus calculator

SUMMARY:
The investigators hypothesize that non-optimally treated carbohydrate counting-naïve patients with type 1 diabetes can achieve better metabolic control by counting carbohydrates and that the metabolic control can be further improved with concurrent use of an integrated glucose meter and bolus calculator. The investigators want to test the hypothesis in this study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Diabetes duration at least 12 months
* MDI therapy
* HbA1c 8-10,5% (both included)

Exclusion Criteria:

* Gastroparesis
* Present or former practice of carbohydrate counting
* Pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 4 months

SECONDARY OUTCOMES:
Variation in blood glucose | 4 months
  Measured by CGM
Number of hypoglycemic events | 4 months
  BG < or = 2.8 and/or unconsciousness
Treatment satisfaction | 4 months
  Questionnaires
Total daily insulin dose | 4 months
Weight | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Signe Schmidt, MD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Schmidt S, Meldgaard M, Serifovski N, Storm C, Christensen TM, Gade-Rasmussen B, Norgaard K. Use of an automated bolus calculator in MDI-treated type 1 diabetes: the BolusCal Study, a randomized controlled pilot study. Diabetes Care. 2012 May;35(5):984-90. doi: 10.2337/dc11-2044. Epub 2012 Feb 16. PMID 22344610